CLINICAL TRIAL: NCT02625168
Title: Efficacy and Safety of Afatinib in Patients With EGFR-mutated Metastatic Non-small-cell Lung Cancer Previously Responsive to First-generation Tyrosine-kinase Inhibitors and Chemotherapy
Brief Title: Afatinib vs Erlotinib as 2nd TKI After Failure to 1st TKI and Chemotherapy for Metastatic NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Victor H.F. Lee, Clinical Assistant Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 1
Record Dates: First submitted 2015-12-02; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Lung Cancer
Keywords: Afatinib; Erlotinib; Metastatic non-small cell lung cancer; Efficacy; Safety
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Afatinib (Experimental): Afatinib 30 or 40 or 50mg daily orally after study recruitment until radiologically documented disease progression, intolerable side effects as judged by investigators or patient withdrawal.
  Interventions: Drug: Afatinib; Drug: Erlotinib
- Erlotinib (Experimental): Erlotinib 150mg daily until radiologically documented disease progression, intolerable side effects as judged by investigators or patient withdrawal.
  Interventions: Drug: Afatinib; Drug: Erlotinib

INTERVENTIONS:
Drug: Afatinib — Afatinib from study recruitment until disease progression, intolerable side effects as judged by investigators or patient withdrawal
  Other Names: Gilotrif
Drug: Erlotinib — Erlotinib from study recruitment until disease progression, intolerable side effects as judged by investigators or patient withdrawal
  Other Names: Tarceva

SUMMARY:
The investigators prospectively evaluated in this study the efficacy and safety profiles of afatinib as 3rd or 4th line treatment after prior failure to systemic chemotherapy and first-generation EGFR-TKI under a Boehringer Ingelheim sponsored Compassionate Use Program (CUP), with comparison of our historical cohort who received erlotinib after previous failure to systemic chemotherapy and first-generation EGFR-TKI.

DETAILED DESCRIPTION:
Study background The investigators prospectively evaluated the use of afatinib as 3rd or 4th line treatment after progression to one line of first-generation EGFR-TKI therapy and at least one line of systemic chemotherapy under this CUP. All patients had documented EGFR activating mutations before the start of afatinib. Determination of EGFR mutation analysis of all patients was described previously. Formalin-fixed paraffin-embedded tumor biopsies before starting 1st TKI therapy were retrieved. Briefly, tumor enrichment was performed by micro-dissection under light microscopy. Genomic DNA was extracted using QIAmp DNA FFPE Tissue kit (Qiagen, Hilden, Germany), followed by polymerase chain reaction (PCR) amplification of EGFR exons 18 to 21 using intron-based primers and sequenced in both forward and reverse directions.

Study population Patients who had EGFR-mutated metastatic NSCLC with prior documented objective response to first-generation TKI (gefitinib or erlotinib) for 6 months and prior treatment of at least 1 line of systemic chemotherapy were eligible to join the CUP offered by Boehringer-Ingelheim Pharma GmbH, Ingelheim, Germany. Patients who had received anti-vascular endothelial growth factor antagonist but not anti-EGFR monoclonal antibody in their previous courses of treatment, either alone or in combination with systemic chemotherapy were allowed to join this CUP. They all had baseline computed tomography scan of the brain, thorax and abdomen with at least 1 evaluable lesion and adequate serum hematological, hepatic and renal function as defined by LUX-Lung1 study.

Treatment The treating physicians then decided the starting dose of afatinib of either 50 mg, 40 mg or 30 mg once daily continuously. After commencement of afatinib, they had regular clinical follow up every 2 weeks for 4 weeks then every 4 weeks until permanent discontinuation of afatinib or death. They also had regular imaging with CT scan every 8-10 weeks for tumor response evaluation by Response Evaluation Criteria for Solid Tumors (RECIST) version 1.1 [16]. Treatment interruption was needed for those who developed grade >= 3 adverse event until it was returned to grade 1 or less. Then afatinib could be resumed but at a one lower dose level. Those who received afatinib 30 mg daily as the initial starting dose would discontinue afatinib permanently if they developed grade >=3 events.

Assessment of efficacy and treatment-related toxicities All treatment-related toxicities were collected and graded according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Objective response (OR) included complete response and partial response while disease control (DC) included complete response, partial response and stable disease according to RECIST 1.1. Survival outcomes included progression-free survival (PFS, defined as time from start of afatinib to first of date of objectively determined progressive disease or death from any cause) and overall survival (OS, time from start of afatinib to date of death from any cause). Time to progression (TTP) started from the date of afatinib commencement to the date of objectively determined progressive disease. All these parameters in those who received afatinib in this study were compared to a historical cohort of patients who received erlotinib after prior failure to gefitinib and at least one line of systemic chemotherapy. All patients in the historical cohort received erlotinib at 150 mg once daily, with the same treatment response evaluation, survival and toxicity assessment as for those who received afatinib.

Statistical analysis Mann-Whitney U was used for comparison of non-parametric variables and chi-square tests were performed for discrete variables. Kaplan-Meier methods with log-rank tests were employed for comparison of survival outcomes and Cox proportional hazard models were used for prognostic factors for PFS after afatinib or erlotinib in univariate and multivariate analyses, with afatinib versus erlotinib, age, sex, performance status, smoking status, histology, TTP for 1st TKI therapy, time interval between 1st TKI and afatinib or erlotinib, TTP for all lines of prior chemotherapy, time interval between last chemotherapy and afatinib or erlotinib as covariates. All statistical analyses were performed by Statistical Package for Social Sciences (SPSS) version 20.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stage IV epidermal growth factor receptor (EGFR)-mutated non-small cell lung cancer who were previously responsive to one line of EGFR tyrosine kinase inhibitor and at least one line of systemic chemotherapy
* Adequate hematological function (ANC >=1.5 x 10^9/l, Hb >=9.0 x 10^9/l, plt >=100 x 10^9/l)
* Adequate renal function (with estimated creatinine clearance >=50ml/min as determined by Cockcroft-Gault formula)
* Adequate liver function (ALT/AST <2.5 x upper normal limit or ALT/AST <5 x upper normal limit in the presence of liver metastasis)
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
* Evaluable target lesions according to RECIST 1.1 for tumour response assessment
* Patients able to give written consent

Exclusion Criteria:

* Symptomatic brain metastases requiring steroids/surgery/radiation therapy within 4 weeks of commencement of study medication
* Significant cardiovascular abnormalities
* Significant psychiatric disorders
* Patients who have documented history of interstitial lung disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From date of start of study medication until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Time interval between date of start of afatinib or erlotinib to date of disease progression or death whichever comes earlier

SECONDARY OUTCOMES:
Objective response rate | Through study completion, an average of 12 months
  Percentage of patients who derive objective response after drug treatment as judged by RECIST 1.1
Overall survival | From date of start of study medication until the date of death from any cause, assessed up to 100 months
  Time interval between date of start of afatinib/erlotinib and date of death from any cause
Toxicity profiles | Through study completion, an average of 12 months
  Adverse events or serious adverse events after afatinib/erlotinib

CONTACTS AND LOCATIONS:
Overall Officials: Victor Lee, MD, Principal Investigator — Department of Clinical Oncology, The University of Hong Kong
Locations (1):
- Department of Clinical Oncology, Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Lee VH, Leung DK, Choy TS, Lam KO, Lam PM, Leung TW, Kwong DL. Efficacy and safety of afatinib in Chinese patients with EGFR-mutated metastatic non-small-cell lung cancer (NSCLC) previously responsive to first-generation tyrosine-kinase inhibitors (TKI) and chemotherapy: comparison with historical cohort using erlotinib. BMC Cancer. 2016 Feb 24;16:147. doi: 10.1186/s12885-016-2201-9. PMID 26911310